CLINICAL TRIAL: NCT02814539
Title: Brain Network Function in School-age Children With Congenital Heart Disease and Its Relation to Higher Order Cognitive Functions
Brief Title: Brain Function in Children With Congenital Heart Disease (CHD)
Status: Completed | Type: Observational
Sponsor: Bea Latal (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor-Investigator, Bea Latal, Prof Dr med Bea Latal, University Children's Hospital, Zurich
Organization: University Children's Hospital, Zurich (Other)
Other Study IDs: BF_CHD_1
Record Dates: First submitted 2016-06-23; First posted 2016-06-27 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- congenital heart disease: children with severe congenital heart disease who undergo open heart surgery during infancy
- healthy controls

SUMMARY:
The purpose of the study is to determine whether the neurodevelopmental outcome and in particular executive functions in 9 to 14 year old school children with congenital heart disease who underwent cardiopulmonary bypass surgery during their first three months of life is impaired in comparison to healthy children at same age. Executive functions are higher order cognitive functions and critical for school success.

ELIGIBILITY:
Inclusion Criteria:

* Congenital heart disease,
* Cardiopulmonary bypass surgery during first three months of life,
* No genetic syndrome,
* Gestational age > 37 weeks of gestation.

Exclusion Criteria:

* Heart surgery without cardiopulmonary bypass,
* Heart surgery not within first three months of life,
* Born <37 weeks of gestation,
* Any genetic syndrome detected.

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-03; Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Executive Functions, assessed with D-KEFS | 2 years

SECONDARY OUTCOMES:
slow wave activity on EEG | 2 years
MRI volumetry | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bea Latal, MD MPH, Principal Investigator — University Childrens Hospital Zurich

IPD SHARING:
Plan to Share IPD: Undecided